CLINICAL TRIAL: NCT02025738
Title: Perioperative MAnaGement of patieNts With Cardiac Implantable Electronic Devices: Randomized Controlled Pilot Trial (MAGNET Trial)
Brief Title: Perioperative Management of Patients With Cardiac Implantable Electronic Devices
Acronym: MAGNET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Mahmoud Suleiman MD, MD, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAGNET2014
Record Dates: First submitted 2013-12-24; First posted 2014-01-01 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: CARDIAC PACEMAKERS DEFIBRILLATOR ELECTROMAGNETIC

ARMS (3):
- MAGNET (Active Comparator): magnet application over cardiac device
  Interventions: Device: MAGNET APPLICATION
- REPROGRAMING (Active Comparator): reprograming of cardiac device by trained technician/electrophysiologist
  Interventions: Device: REPROGRAMING
- NO ACTION (Active Comparator): no action is performed if patient meets inclusion criteria
  Interventions: Device: NO ACTION

INTERVENTIONS:
Device: MAGNET APPLICATION
  Arms: MAGNET
Device: REPROGRAMING
  Arms: REPROGRAMING
Device: NO ACTION
  Arms: NO ACTION

SUMMARY:
Data on the perioperative management of patients cardiac implantable electronic devices (CIEDs) is limited and published guidelines rely mainly on the experience of the cardiologists and anesthesiologists who manage these patients. Depending on the device type and patient's dependency, these guidelines recommend the intraoperative magnet use, reprogramming of devices or no action. Magnet placement on a CIED (very simple and applicable method) has become the standard approach in many centers, while CIED reprograming by trained personnel is required in most centers. Therefore, our objective is to compare in a prospective randomized clinical trial the safety of intraoperative magnet use vs. CIEDS reprogramming vs. no intervention (in the appropriate subjects)

ELIGIBILITY:
Inclusion Criteria:

* All subjects with cardiac implanted electronic device (CIED) who are candidates of non-cardio-thoracic surgery or endoscopy and anticipated use of electrocautery

Exclusion Criteria:

* Recent CIED implantation (less than 6 weeks)
* Subjects with ICD who are pacemaker dependent
* Cardio - thoracic surgery
* Surgery over the CIED site
* Surgery site that preclude use of magnet in efficient way
* Subjects with Implanted unipolar leads

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Any inappropriate sensing of EMI caused by electrocautery. | DURING SURGERY/PROCEDURE

SECONDARY OUTCOMES:
Any significant change in CIEDS parameters | WITHIN 1 DAY OF SURGERY/PROCEDURE

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Medical Center, Haifa, Israel

REFERENCES:
- [Background] Crossley GH, Poole JE, Rozner MA, Asirvatham SJ, Cheng A, Chung MK, Ferguson TB Jr, Gallagher JD, Gold MR, Hoyt RH, Irefin S, Kusumoto FM, Moorman LP, Thompson A. The Heart Rhythm Society (HRS)/American Society of Anesthesiologists (ASA) Expert Consensus Statement on the perioperative management of patients with implantable defibrillators, pacemakers and arrhythmia monitors: facilities and patient management this document was developed as a joint project with the American Society of Anesthesiologists (ASA), and in collaboration with the American Heart Association (AHA), and the Society of Thoracic Surgeons (STS). Heart Rhythm. 2011 Jul;8(7):1114-54. doi: 10.1016/j.hrthm.2010.12.023. No abstract available. PMID 21722856